CLINICAL TRIAL: NCT02305251
Title: Patient Preferences of a Resect and Discard Paradigm
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Dayna Early, Professor of Medicine, Washington University School of Medicine
Other Study IDs: 201202031
Record Dates: First submitted 2014-11-19; First posted 2014-12-02 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Survey — Standard Gamble Survey

SUMMARY:
The investigators conducted a study "Resect and Discard Diminutive Polyps: a new paradigm" (IRB ID # 201105473) from September, 2011 to July, 2013. This study examined whether doctors performing colonoscopy are accurate enough at predicting histology of small colorectal polyps, such that these small polyps could be resected and discarded (instead of being sent to pathology). One of the main advantages of this approach is significant cost savings by reducing pathology costs associated with screening and surveillance colonoscopy. A disadvantage is that there is a 0.03% chance that small polyps contain cancer. There is no data regarding patient preferences toward this approach. The investigators therefore designed a patient survey to determine the patient's view toward this approach.

DETAILED DESCRIPTION:
The American Society of Gastrointestinal Endoscopy (ASGE) published a review article on a new paradigm in colorectal cancer screening termed "resect and discard". This new paradigm challenges the current practice of sending all colorectal polyps, regardless of appearance or size, to pathology for analysis. "Resect and Discard" describes a new approach in which small polyps could be removed, but be discarded instead of sent for pathology analysis. This is based on data showing that gastroenterologists can predict the pathology of small colorectal polyps with 80-90% accuracy, and that discarding small polyps would not alter surveillance recommendations.

Neither the ASGE document nor published research, however, assessed patient attitudes toward this approach. This study surveyed patients prior to first time screening colonoscopy, in order to determine their preferences about the resect and discard approach; specifically would patients be willing to pay for pathology analysis of small colorectal polyps with their own money, and what factors influence their decision. We also inquired about factors that would influence their decision to pay/not pay pathology costs themselves.

ELIGIBILITY:
Inclusion Criteria:

• Indication for colonoscopy is screening or routine polyp surveillance

Exclusion Criteria:

* Indication for colonoscopy other than screening or surveillance
* Colon cancer identified at time of colonoscopy
* Known polyposis syndrome, or polyposis identified at colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients reporting in for colonoscopies either for screening or for polyp surveillance.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2015-11-02 (Actual)

PRIMARY OUTCOMES:
Number of participants willing to pay out of pocket for pathology costs when a diminutive polyp is found. | June, 2012 to March, 2014: up to 2 years
  This outcome is measured in percentage.

SECONDARY OUTCOMES:
The factors that influence patients' decisions to pay or not pay for pathology costs with their own money. | June, 2012 to March, 2014: up to 2 years
  These factors were measured using univariate analysis with generation of odds ratios and 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Dayna S Early, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Hassan C, Pickhardt PJ, Rex DK. A resect and discard strategy would improve cost-effectiveness of colorectal cancer screening. Clin Gastroenterol Hepatol. 2010 Oct;8(10):865-9, 869.e1-3. doi: 10.1016/j.cgh.2010.05.018. Epub 2010 Jun 1. PMID 20621680
- [Background] Rex DK. Narrow-band imaging without optical magnification for histologic analysis of colorectal polyps. Gastroenterology. 2009 Apr;136(4):1174-81. doi: 10.1053/j.gastro.2008.12.009. Epub 2008 Dec 10. PMID 19187781
- [Derived] Vu HT, Sayuk GS, Gupta N, Hollander T, Kim A, Early DS. Patient preferences of a resect and discard paradigm. Gastrointest Endosc. 2015 Aug;82(2):381-384.e1. doi: 10.1016/j.gie.2015.01.042. Epub 2015 Apr 22. PMID 25910663